CLINICAL TRIAL: NCT01071707
Title: COMET: Correlating Outcomes With Biochemical Markers to Estimate Time-progression in IPF. A Prospective, Multi-Center, Longitudinal Follow up Study of Subjects With Idiopathic Pulmonary Fibrosis
Brief Title: Correlating Outcomes With Biochemical Markers to Estimate Time-progression in Idiopathic Pulmonary Fibrosis (IPF)
Acronym: COMET
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Fernando J. Martinez, MD, MS, University of Michigan
Other Study IDs: COMET; 1RC2HL101740-01 (NIH)
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2009-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: IPF; Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Confirmed Diagnosis of IPF: Subjects in this cohort will continue beyond the screening visit(s) for longitudinal follow up visits for a minimum of 48 weeks and maximum of 80 weeks.
- No diagnosis of IPF: Subjects that complete screening visits and do not obtain a confirmed diagnosis of IPF will conclude the study at screening, at the time point where IPF is ruled out as a diagnosis.

SUMMARY:
Study purpose:

The disease course of idiopathic pulmonary fibrosis (IPF) is variable. During the course of the disease some patients will get better, some will stay the same, and others will get worse. Currently doctors do not have any way to predict an individual patients disease course. The purpose of this study is to determine if 'biomarkers' such as proteins or genes isolated at the time of diagnosis can be used to predict the disease course. These 'biomarkers' will be obtained from samples of blood, from a procedure call a bronchoscopy, and in some patients from extra tissue obtained by a surgical lung biopsy.

DETAILED DESCRIPTION:
The objectives of this study are as follows:

Specific Aim 1: Assemble a network of clinical centers to procure biologic samples from subjects with recently diagnosed IPF and follow these subjects for at least 48 weeks. Specific Aim 2: Correlate and integrate biologically plausible biomarkers of disease activity obtained from multiple compartments (SLB, BAL, TBB, blood) from the same subject with longitudinal measures of disease progression (change in forced vital capacity, change in diffusion capacity for carbon monoxide, acute exacerbation of pulmonary fibrosis, and death).

General Study Design This study will take place in two phases. During the first phase of the study we will identify and collect baseline specimens from subjects with either suspected or recently diagnosed (within 48 months) IPF. During the second phase of the study subjects with IPF will be followed from between 48 and 80 weeks. Subjects will be followed until the end of study (2 year grant award) or until they meet any part of a composite endpoint (death, acute exacerbation of IPF, relative decline in FVC of at least 10% or DLCO of 15%). This is a prospective cohort study. There is no treatment prescribed or studied as part of this prospective cohort study. Subjects are able to utilize any treatments prescribed by their physician, including participation in clinical trials as long as they are able to comply with the follow up schedule in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected or confirmed diagnosis of IPF
2. Age 35 - 80 years inclusive
3. Ability to understand and provide informed consent

Exclusion Criteria:

1. Confirmed diagnosis of IPF at the study center more than 4 years prior to screening
2. Environmental exposure (occupational, environmental, drug, etc) felt by the principal investigator (PI) to be the etiology of the interstitial disease
3. Diagnosis of collagen-vascular conditions (according to the published American College of Rheumatology criteria)
4. Forced expiratory volume in 1 second (FEV1)/FVC ratio < 0.60 at screening (postbronchodilator)
5. Significant bronchodilator response on screening spirometry, defined as a change in FEV1 ≥ 12% and absolute change > 200 mL OR change in FVC ≥ 12% and absolute change > 200 mL
6. Evidence of active infection at screening
7. Listed for lung transplantation at time of screening
8. Unstable or deteriorating cardiac disease at screening
9. Myocardial infarction, coronary artery bypass, or angioplasty within 6 months of screening
10. Unstable angina pectoris or congestive heart failure requiring hospitalization within 6 months of screening
11. Uncontrolled arrhythmia at screening
12. Severe uncontrolled hypertension at screening
13. Known HIV or hepatitis C at screening
14. Known cirrhosis or chronic active hepatitis at screening
15. Active substance and/or alcohol abuse at screening
16. Subjects who are pregnant or breastfeeding at screening
17. Women of childbearing potential who are not using a medically approved means of contraception at screening
18. Known bleeding abnormality that would preclude the performance of transbronchial lung biopsy
19. Prothrombin time, INR > 1.5, Partial Thromboplastin Time (PTT) > 45 at time of screening, platelets < 100,000/mm3
20. Any condition other than IPF that, in the opinion of the site PI, is likely to result in the death of the subject within the next year
21. Any condition that, in the judgment of the site PI, might cause participation in this study to be detrimental to the subject or that the site PI deems makes the subject a poor candidate

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with suspected or confirmed diagnosis of Idiopathic Pulmonary Fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2009-12; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome is progression free survival as determined by time until any of: death, acute exacerbation of IPF, relative change in FVC (liters) of at least 10% or DLCO (ml/min/mmHg) of 15%. | Follow up visits after baseline, every 16 weeks for minimum of 40 weeks and maximum of 80 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Reynolds, MD, Study Director — National Heart, Lung and Blood Institute, Division of Lung Sciences, National Institute of Health; Fernando J Martinez, MD,MS, Principal Investigator — University of Michigan; Galen B Toews, MD, Principal Investigator — University of Michigan; Kevin R Flaherty, MD, MS, Principal Investigator — University of Michigan
Locations (9):
- United States (9):
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - University of Chicago, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Temple University, Philadelphia, Pennsylvania
  - Brown University, Providence, Rhode Island
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Derived] Allen RJ, Stockwell A, Oldham JM, Guillen-Guio B, Schwartz DA, Maher TM, Flores C, Noth I, Yaspan BL, Jenkins RG, Wain LV; International IPF Genetics Consortium. Genome-wide association study across five cohorts identifies five novel loci associated with idiopathic pulmonary fibrosis. Thorax. 2022 Aug;77(8):829-833. doi: 10.1136/thoraxjnl-2021-218577. Epub 2022 Jun 10. PMID 35688625
- [Derived] Whalen W, Buyukozkan M, Moore B, Moon JS, Dela Cruz CS, Martinez FJ, Choi AMK, Krumsiek J, Stout-Delgado H, Cho SJ. Association of circulating cell-free double-stranded DNA and metabolic derangements in idiopathic pulmonary fibrosis. Thorax. 2022 Feb;77(2):186-190. doi: 10.1136/thoraxjnl-2021-217315. Epub 2021 Sep 14. PMID 34521729
- [Derived] Galli JA, Panetta NL, Gaeckle N, Martinez FJ, Moore B, Moore T, Courey A, Flaherty K, Criner GJ; COMET investigators. Pneumothorax After Transbronchial Biopsy in Pulmonary Fibrosis: Lessons from the Multicenter COMET Trial. Lung. 2017 Oct;195(5):537-543. doi: 10.1007/s00408-017-0028-z. Epub 2017 Jun 16. PMID 28623539
- [Derived] Han MK, Zhou Y, Murray S, Tayob N, Noth I, Lama VN, Moore BB, White ES, Flaherty KR, Huffnagle GB, Martinez FJ; COMET Investigators. Lung microbiome and disease progression in idiopathic pulmonary fibrosis: an analysis of the COMET study. Lancet Respir Med. 2014 Jul;2(7):548-56. doi: 10.1016/S2213-2600(14)70069-4. Epub 2014 Apr 21. PMID 24767767